CLINICAL TRIAL: NCT00838890
Title: A Phase 1/2, Multiple Ascending Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-863233 in Subjects With Refractory Hematologic Malignancies
Brief Title: A Study of BMS-863233 in Patients With Hematologic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA198-001
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Refractory Hematologic Cancer
MeSH Terms: conditions — Hematologic Neoplasms

ARMS (2):
- Cdc7-inhibitor (A) (Active Comparator)
  Interventions: Drug: Cdc7-inhibitor (BMS-863233)
- Cdc7-inhibitor (B) (Active Comparator)
  Interventions: Drug: Cdc7-inhibitor (BMS-863233)

INTERVENTIONS:
Drug: Cdc7-inhibitor (BMS-863233) — Tablets, Oral, QD x 14 days until MTD is achieved, 14 days per 28 day cycle/QD, 12 months
  Other Names: BMS-863233
  Arms: Cdc7-inhibitor (A)
Drug: Cdc7-inhibitor (BMS-863233) — Tablets, Oral, MTD of Cdc7-inhibitor (A) Arm, QD x 7 days until MTD achieved, 7 days per 21 day cycle/QD, 12 months
  Other Names: BMS-863233
  Arms: Cdc7-inhibitor (B)

SUMMARY:
To determine safety, tolerability and maximum tolerated dose of BMS-63233/XL413 in subjects with Refractory Hematologic Cancer

ELIGIBILITY:
Inclusion Criteria:

* AML by current WHO diagnostic criteria, any FAB type (except APML), Refractory ALL, Accelerated/blast phase CML and Refractory MDS with total IPSS score of 2 or higher
* ECOG performance status <= 2
* Accessible for treatment, PK sample collection and required study follow-up
* Total Bilirubin ≤ 1.5 x ULN and ALT, AST ≤ 3 x ULN

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Subjects with Acute Promyelocytic leukemia disease or CNS leukemia disease)
* Hyperleukocytosis (defined as peripheral WBC >50,000/uL)
* Treatment with any other investigational agent for any indication within 30 days of protocol enrollment
* Subjects a history of gastrointestinal disease
* Subjects less than four weeks from allogenic or autologous stem cell transplant infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine maximum tolerated dose and anti-tumor activity of BMS-863233/XL413 when administered to subjects with refractory Hematologic Cancer | Every 21 or 28 days until maximum tolerated dose is reached

SECONDARY OUTCOMES:
To determine the safety of BMS-863233/XL413 when administered to subjects with refractory Hematologic Cancer | Every 21 or 28 days until the MTD is reached
To determine the pharmacokinetics of BMS-863233/XL413 when administered to subjects with refractory Hematologic Cancer | Every 21 or 28 days until the MTD is reached
To determine the anti-tumor activity of BMS-863233/XL413 when administered to subjects with refractory Hematologic Cancer | Every 21 or 28 days until the MTD is reached

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - University Of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Roswell Park, Buffalo, New York

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx